CLINICAL TRIAL: NCT04415268
Title: Combined Effect of CFTR Protein Modulator Drugs and Exercise on Pulmonary Function, Fitness, Sweat Test and Quality of Life in Children With Cystic Fibrosis
Brief Title: Combined Effect of CFTR Protein Modulator Drugs and Exercise in Cystic Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we did not receive expected funding
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Full Professor MD, PhD, Universidad Europea de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIPI/20/119
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Electrostimulation; Combined Training; Physical Fitness
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-group non-randomized, prospective. Within-subject multitreatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multitreatment (Experimental): Pharmacological treatment per standard of care (whole study length, starting on week 1).
  Supervised exercise protocol (phase 1, 8 weeks starting on week 9). Unsupervised exercise protocol (phase 2, 8 weeks starting on week 17).
  Interventions: Behavioral: Exercise; Behavioral: Unsupervised exercise; Drug: CFTR Modulators

INTERVENTIONS:
Behavioral: Exercise — Surpervised exercise program: Includes a concurrent exercise intervention (strength training and aerobic training), 3 days a week, 60 minutes sessions.
Behavioral: Unsupervised exercise — Unsupervised exercise program: The same exercise program learned during the supervised phase will be practiced at home.
Drug: CFTR Modulators — Standard of care: Lumacaftor with Ivacaftor or Tezacaftor combined with Ivacaftor.
  For children between 6 and 11 years of age, Lumacaftor 400 mg combined with Ivacaftor 500 mg in total per day, divided into 2 doses per day; for those over 11 years of age, Tezacaftor 100 mg combined with Ivacaftor 150 mg in the morning, adding a dose of Ivacaftor 150 mg at night.
  https://www.clinicaltrialsregister.eu/ctr-search/trial/2019-000833-37/ES
  Other Names: EudraCT Number 2019-000833-37

SUMMARY:
This study aims to assess the effects of programmed exercise combined with CFTR protein modulator drugs in the cardiorespiratory fitness, strength, functional capacity and agility in a group of young patients with Cystic Fibrosis.

DETAILED DESCRIPTION:
The present study is a new clinical trial that extends our previous work intended to assess the effect of programmed exercise with or without electrical stimulation on cardiorespiratory fitness, strength, functional capacity and agility in a group of young patients with Cystic Fibrosis (ECOMIRIN) registered at ClinicalTrials.gov (Identifier: NCT04153669).

After finishing the study, a subset of the participants was treated with either TEZ/IVA or LUM/IVA per standard of care, as they were considered candidates according to the AEMPS (https://www.clinicaltrialsregister.eu/ctr-search/trial/2019-000833-37/ES). Those patients are expected to complete five months of pharmacological treatment without exercise by June 2020.

Primary Objective To evaluate the effect of an exercise program on physical fitness in cystic fibrosis patients after 5 months of administration of LUM/IVA or TEZ/IVA in comparison to the effect produced by the same exercise program before administration of the drug.

Secondary Objectives Other specific objectives include comparing the beneficial effects of exercise and LUM/IVA or TEZ/IVA on: 1) cardiorespiratory function and muscle strength; 2) the concentration of chlorine in sweat; and 3) quality of life.

ELIGIBILITY:
Inclusion Criteria:

* In order to be included, patients must have participated in the ECOMIRIN clinical trial (ClinicalTrials.gov Identifier: NCT04153669).
* They must have a previous CF diagnosis, defined as: sweat chlorine ≥ 60 mEq/L and/or carry two variants of the CFTR gene characterized as pathogenic.
* Age 6-18 years; eligible to receive treatment with TEZ/IVA or LUM/IVA according to the AEMPS (LUM/IVA for 6-11 year-old children homozygous for the F508del mutation; TEZ/IVA for ≥ 12 year-old children homozygous for the Phe508del mutation, as well as heterozygous for the F508 mutation plus one of the following mutations: P67L, R117C, L206W, R352Q, A455E, D579G, 711 + 3A G, S945L, S977F, R1070W, D1152H, 2789 + 5G A, 3272-26A G, and 3849 + 10kbC T);
* Agreement to collaborate in performing static and dynamic pulmonary function tests.
* Consent of children and/or parents or legal guardians to participate in the study after having read and understood the informed consent form.

Exclusion Criteria:

* CF patients not consenting to participate in the study at any time after reading and understanding the informed consent form will be excluded.
* CF patients who are not eligible to receive treatment with TEZ/IVA or LUM/IVA according to the AEMPS during the course of the study will be excluded.
* Study participants will be excluded if they test positive for any contagious viral infection that may affect the outcomes (e.g. SARS-CoV-2).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-09 (Estimated); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in Strength | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in strength will be measured using a five repetition maximum test (5RM)
Change in Cardiorespiratory Fitness | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in cardiorespiratory fitness will be measured using a cardiopulmonary exercise test (CPET)

SECONDARY OUTCOMES:
Changes in Forced expiratory volume in 1 second (FEV1) | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in FEV1 will be measured using Spirometry (z-score based on Global Lung Function Initiative reference DOI: 10.1016/j.arbres.2017.07.019)
Changes in Forced vital capacity (FVC) | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in FVC will be measured using Spirometry (z-score based on Global Lung Function Initiative reference DOI: 10.1016/j.arbres.2017.07.019)
Changes in FEV1/FVC ratio (FEV1%) | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in FEV1/FVC ratio (FEV1%) will be measured using Spirometry (z-score based on Global Lung Function Initiative reference DOI: 10.1016/j.arbres.2017.07.019)
Changes in Forced expiratory flow (FEF) | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in FEF will be measured using Spirometry (z-score based on Global Lung Function Initiative reference DOI: 10.1016/j.arbres.2017.07.019)
Changes in Physical Activity Questionnaire (PAQ) for children and adolescents | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in physical activity levels will be measured using PAQ-C for children under 14 years of age and PAQ-A for adolescents over 14 years of age.
  Items 1 to 9 will be used in the physical activity composite score, and means will be calculated to obtain the final PAQ-C activity summary score. Items 1 to 8 will be used in the physical activity composite score, and means will be calculated to obtain the final PAQ-A activity summary score.
  A score of 1 indicates low physical activity, whereas a score of 5 indicates high physical activity.
Change in quality of life: Cystic Fibrosis-Questionnaire-Revised (CFQ-R) | Four assessment points throughout the study: baseline and after each 8-week intervention
  Changes in quality of life will be measures with the Cystic Fibrosis-Questionnaire-Revised (CFQ-R).
  Scores for each health related quality of life domain are calculated; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health.
Sweat chloride level | Four assessment points throughout the study: baseline and after each 8-week intervention
  Chloride concentration in sweat (mEq/L) will be measured in the laboratory using an MK II Chloride Analyzer 926S

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez-Ruiz, MD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Escuela de Doctorado e Investigacion, Universidad Europea, Villaviciosa de Odón, Spain